CLINICAL TRIAL: NCT03910712
Title: A Randomized, Open-label Study of First Line Pyrotinib, Trastuzumab With an Aromatase Inhibitors, in the Treatment of HER2 Positive and HR Positive Metastatic or Inoperable Locally Advanced Breast Cancer
Brief Title: Pyrotinib Combined With Trastuzumab and AI in the First-line Treatment of HER2 Positive/ HR Positive MBC
Acronym: Pyrotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiang SUN, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREAST-Pyrotinib
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer Female; HER2-positive Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; Metastatic Breast Cancer; Breast Diseases; Hormone Receptor Positive Tumor
Keywords: MBC, Pyrotinib, Trastuzumab, First line, HER2
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — pyrotinib; Drug Evaluation; Trastuzumab; Aromatase Inhibitors; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrotinib and trastuzumab plus aromatase inhibitor (Experimental): Participants will receive pyrotinib in combination with trastuzumab plus AI until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Aromatase inhibitor
- Trastuzumab plus aromatase inhibitor (Active Comparator): Participants will receive trastuzumab plus AI until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Trastuzumab; Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib were administered 400 mg orally daily. Oral administration within 30 minutes after breakfast, and continuous administration for 21 days for 1 cycle.
  Other Names: Study drug
  Arms: Pyrotinib and trastuzumab plus aromatase inhibitor
Drug: Trastuzumab — Trastuzumab were administered every 3 weeks intravenously (8 mg/kg loading doses followed by 6 mg/kg maintenance doses).
  Other Names: Herceptin®
Drug: Aromatase inhibitor — The investigator chose an aromatase inhibitor (either anastrozole, letrozole or exemestane 1 mg/2.5 mg/25 mg), once daily, oral.
  Other Names: anastrozole, letrozole or exemestane

SUMMARY:
This study is a randomized, open-label, phase II study, comparing the efficacy and safety of trastuzumab plus aromatase inhibitors, with or without pyrotinib, in the treatment of HR (hormone receptor)+/HER2 (human epidermal growth factor receptor 2) + MBC and inoperable LABC patients.

DETAILED DESCRIPTION:
This is a randomized, two-arm, open-label, multicenter phase II trial. Our primary purpose is to compare that PFS of patients with trastuzumab, AI plus pyrotinib and trastuzumab plus an AI for HER2-positive and hormone receptor-positive MBC or locally advanced breast cancer (LABC).

Eligible patients will randomized to a ratio of 1:1 to pyrotinib+ trastuzumab + aromatase inhibitor (experimental group) or trastuzumab+aromatase inhibitor (control group). Stratification factors were 1)time since adjuvant hormone therapy (<=12 months/>12 months/no prior hormone therapy); 2) lesion (visceral; non-visceral).

In treatment period, patients will be administrated trastuzumab plus aromatase inhibitors, with or without pyrotinib, every 21 days for 1 cycle, until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, female;
2. Postmenopausal or pre-menopausal with ovarian function suppression;
3. At least one measurable lesion evaluable according to Response Evaluation Criteria In Solid Tumors Version 1.1;
4. Metastatic or inoperable local advanced breast cancer;
5. HER2-positive breast cancer;
6. HR-positive breast cancer;
7. LVEF ≥50%;

Exclusion Criteria:

1. Previous systemic non-hormonal anticancer therapy in the metastatic or advanced breast cancer setting;
2. Received endocrine therapy within 7 days before randomization;
3. Uncontrolled central nervous system metastases;
4. Disease-free interval from completion of adjuvant/neo-adjuvant systemic non-hormonal treatment to recurrence of within 6 months.
5. Other malignancies within the last 3 years, except for carcinoma in situ of the cervix or basal cell carcinoma.
6. Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during the course of study treatment
7. Severe organ dysfunction as assessed by signs and symptoms, laboratory studies and rapid progression of disease, which leading to a clinical indication for chemotherapy.
8. History of CHF of any New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (exception, atrial fibrillation, paroxysmal supraventricular tachycardia);
9. History of myocardial infarction within 6 months of randomization
10. History of LVEF decline to below 50% during or after prior trastuzumab neo-adjuvant or adjuvant therapy
11. Pregnant or lactating women;
12. QT interval>470 ms；
13. Serious concomitant diseases (including severe hypertension, severe diabetes, active infection, thyroid disease, etc.) that are harmful to the patient's safety or affect the patient's completion of the study;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to 36 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization to 36 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Objective Overall Response Rate (ORR) | From randomization to 36 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Duration of Response (DoR) | From randomization to 36 month
  DoR is defined as date of initial confirmed PR/CR until date of progressive disease or death from any cause. PR or CR or SD is according to RECIST version 1.1.
  The DoR will be estimated using Kaplan-Meier method. Kaplan-Meier curves, median DoR, hazard ratio with appropriate confidence intervals will be reported.
Time to Response (TTR) | From randomization to 36 month
  Time to Response (TTR), defined as the time from the date of randomization to the date of first CR or PR. CR or PR is according to RECIST version 1.1.
  The TTR will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median TTR, hazard ratio with appropriate confidence intervals will be reported.
Clinical Benefit Response (CBR) | From randomization to 36 month
  CBR is percentage of participants with best (confirmed) PR or CR or SD for at least 6 months. PR or CR or SD is according to RECIST version 1.1.
  The CBR will be reported by percentage with each arms and appropriate confidence intervals.
Adverse events (AEs) | From screening phase until AEs returns to Grade 0-1 or baseline
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.3.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.
Quality of Life (QoL) by FACT-B | From randomization to 36 month
  QoL was assessed using Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B). FACT-B is a 37-item questionnaire with 5 subscales assessing physical, social, emotional, and functional well-being, as well as a breast cancer specific subscale.
  FACT-B questionnaires were completed by patients on screening phase (baseline) and each 6 weeks after randomization. Mean change from baseline of FACT-B scores by each visit for each arms will be reported.
Quality of Life (QoL) by EQ-5D | From randomization to 36 month
  QoL was assessed using EuroQoL 5-Dimensions (EQ-5D). EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments.
  EQ-5D questionnaires were completed by patients on screening phase (baseline) and each 6 weeks after randomization. Mean change from baseline of EQ-5D scores by each visit for each arms will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, M.D., Study Chair — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Lin Y, Zhou Y, Mao F, Zhu H, Guan J, Zhang X, Shen S, Huang X, Chen C, Yao R, Zhao J, Sun Q. Pyrotinib with trastuzumab and aromatase inhibitors as first-line treatment for HER2 positive and hormone receptor positive metastatic or locally advanced breast cancer: study protocol of a randomized controlled trial. BMC Cancer. 2020 Jul 13;20(1):653. doi: 10.1186/s12885-020-07143-2. PMID 32660609